CLINICAL TRIAL: NCT01531101
Title: First Experimental Study of Transference Work - In Teenagers
Brief Title: First Experimental Study of Transference Work - In Teenagers (FEST-IT)
Acronym: FEST-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randi Ulberg (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor-Investigator, Randi Ulberg, Researcher, Sykehuset i Vestfold HF
Organization: Sykehuset i Vestfold HF (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sykehuset i Vestfold; REK: 2011/1424 FEST-IT (Registry Identifier: The Central Norway Regional Ethics Health Committee)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Depression
Keywords: Transference work; Psychodynamic; Depression; Treatment; Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual PDT with TW (Experimental): Individual Psychodynamic psychotherapy with transference work (TW).
  Interventions: Behavioral: Individual psychodynamic psychotherapy
- Individual PDT without (TW) (Active Comparator): Individual Psychodynamic psychotherapy without focus on transference work (TW).
  Interventions: Behavioral: Individual psychodynamic psychotherapy

INTERVENTIONS:
Behavioral: Individual psychodynamic psychotherapy — Individual psychodynamic psychotherapy with or without transference work. I.e. with or without relational therapist interventions focusing on the patient-therapist relationship.
  Other Names: Individual PDT; Short-term psychodynamic psychotherapy; Short-term dynamic psychotherapy; Short-term psychoanalytic psychotherapy

SUMMARY:
The First Experimental Study on Transference work - In Teenagers (FEST-IT) will be a randomized clinical trial, which will be designed to explore effects of transference work in dynamic psychotherapy in adolescents with major depressive disorder (MDD). The design of the study is a so-called dismantling design, in which a single component is added and/or varied to an existent treatment method (psychodynamic psychotherapy). Thus, the efficiency of a specific technique (transference interventions) can be identified.

The primary hypothesis is that the transference group may have a more favorable course over time than will the comparison group.

The second hypothesis is that patients with a history of low Quality of Object Relations score and/or personality disorders-might benefit more from therapy with transference work than from therapy without.

The third hypothesis is that female adolescents may have better treatment effect of transference work than male adolescents.

DETAILED DESCRIPTION:
The effect of transference interventions in depressed adolescents and the moderator moderating effect of quality of object relations, personality disorder and gender will be explored. Methods and study design: The First Experimental Study of Transference Work-In Teenagers (FEST-IT) will be a randomized clinical trial with a dismantling design. The study is aimed to explore the effects of transference work in psychodynamic psychotherapy for adolescents with depression. One hundred patients ages 16 to 18 years old will be randomized to one of two treatment groups, in both of which general psychodynamic techniques will be used. The quality of adolescents' relationships will be a central focus of the study.The patients will be treated over 28 weeks with either a moderate level of transference intervention or no transference intervention. Follow-up will be at 1 year after treatment termination.

Gender personality disorder (PD) and quality of object relations (QOR) will be the preselected moderators.

The object of this clinical trial is to explore the effect of transference interventions in psychodynamic psychotherapy in adolescents with a major depressive disorder. Using a randomized and dismantling design, we hope that the study will add more specific knowledge to the evidence base.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 16 - 18 years

Exclusion Criteria:

* Pervasive developmental disorder,
* psychosis, or substance abuse

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Psychodynamic Functioning Scales (PFS) | 3 months
  Average of 5 subscales rated by experienced clinician raters; family relations, friendships, tolerance for affects, insight, problem solving and adaptive capacity
Inventory of Interpersonal Problems-Circumplex Version (IIP-C) | Currentl
  64.items patient rated measure

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | One week
  Rated by experienced clinician raters
Symptom Checklist-90 (Global Severity Index; GSI) | Current
  Patient-rated
Beck Depression Inventory (BDI) | Current
  Patient rated
Montgomery Åsberg Rating Scale (MADRS) | Current
  Rated by therapist and/or experienced clinician rater

OTHER OUTCOMES:
Adolescent Relationship Scale (ARS) | Current
  Patient rated Visual-Analogues scales

CONTACTS AND LOCATIONS:
Overall Officials: Randi Ulberg, PhD, Principal Investigator — Vestfold Hospital Trust and University of Oslo
Locations (6):
- Norway (6):
  - Research Unit, Division of, Tønsberg, Vestfold
  - BUP vest, Diakonhjemmet sykehus, Oslo
  - Nic Walls Institutt, Lovisenberg Diakonale Sykehus, Oslo
  - Oslo University Hospital, Oslo
  - Spcialist in psychiatry and clinical psychiatry, Oslo
  - University of Oslo, Oslo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Calderon A, Storeide KAH, Elvejord C, Nissen-Lie HA, Ulberg R, Dahl HJ. Examining Psychotherapeutic Processes with Depressed Adolescents: A Comparative Study of Two Psychodynamic Therapies. Int J Environ Res Public Health. 2022 Dec 16;19(24):16939. doi: 10.3390/ijerph192416939. PMID 36554820
- [Derived] Brosholen P, Ulberg R, Dahl HJ, Thoren A. Therapists' Emotional Responses in Individual Therapy with Depressed Adolescents: An Evaluation of the Data Structure of the Feeling-Word Checklist-28. Int J Environ Res Public Health. 2022 Aug 2;19(15):9496. doi: 10.3390/ijerph19159496. PMID 35954850
- [Derived] Henriksen AK, Ulberg R, Tallberg BPU, Lovgren A, Johnsen Dahl HS. Conflicted Anger as a Central Dynamic in Depression in Adolescents-A Double Case Study. Int J Environ Res Public Health. 2021 Jun 15;18(12):6466. doi: 10.3390/ijerph18126466. PMID 34203924
- [Derived] Ulberg R, Hummelen B, Hersoug AG, Midgley N, Hoglend PA, Dahl HJ. The first experimental study of transference work-in teenagers (FEST-IT): a multicentre, observer- and patient-blind, randomised controlled component study. BMC Psychiatry. 2021 Feb 17;21(1):106. doi: 10.1186/s12888-021-03055-y. PMID 33596856
- [Derived] Lovgren A, Rossberg JI, Nilsen L, Engebretsen E, Ulberg R. How do adolescents with depression experience improvement in psychodynamic psychotherapy? A qualitative study. BMC Psychiatry. 2019 Mar 21;19(1):95. doi: 10.1186/s12888-019-2080-0. PMID 30898111
- [Derived] Ness E, Dahl HJ, Tallberg P, Amlo S, Hoglend P, Thoren A, Egeland J, Ulberg R. Assessment of dynamic change in psychotherapy with asdolescents. Child Adolesc Psychiatry Ment Health. 2018 Jul 30;12:39. doi: 10.1186/s13034-018-0246-z. eCollection 2018. PMID 30069230
- [Derived] Ulberg R, Hersoug AG, Hoglend P. Treatment of adolescents with depression: the effect of transference interventions in a randomized controlled study of dynamic psychotherapy. Trials. 2012 Sep 6;13:159. doi: 10.1186/1745-6215-13-159. PMID 22950546
- See also: The Central Norway Regional Ethics Health Committee — https://helseforskning.etikkom.no/komiteerogmoter/midt/sekretariat?p_dim=34989&region=10797
- See also: Sykehuset i Vesthold — https://www.siv.no/
- See also: University of Oslo — http://www.uio.no
- See also: Ulberg R, Hersoug AG, Høglend P.(2012)Treatment of adolescents with depression: the effect of transference interventions in a randomized controlled study of dynamic psychotherapy.Trials. 2012 Sep 6;13:159. doi: 10.1186/1745-6215-13-159. — http://www.biomedcentral.com/content/pdf/1745-6215-13-159.pdf